CLINICAL TRIAL: NCT01282281
Title: Prospective Metabolic Monitoring of Youth and Adults With Bipolar Disorder.
Status: Completed | Type: Observational
Sponsor: Dr. Ayal Schaffer (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Dr. Ayal Schaffer, Head, Mood & Anxiety Disorders Program; Deputy Psychiatrist-in-Chief, Department of Psychiatry; Associate Professor, University of Toronto, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Other Study IDs: WS688773
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Bipolar Disorder; Youth; Adults
Keywords: Bipolar Disorder; Youth; Adults; Endocrine-metabolic changes
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Individuals aged 14-18 and 19-65 with a diagnosis of BD

SUMMARY:
Background: Most psychotropic medications that are effective in the treatment of Bipolar Disorder (BD) are associated with endocrine-metabolic changes (EMCs). To date, there is no long-term study in BD that has examined specifically the association of inflammation with EMCs in BD. Specific aims: 1) to identify predictors of EMCs among adolescents and adults with BD who are being started on a medication ; 2) to compare change in EMCs in youth and adults treated for BD; 3) to measure change in EMCs associated with use of different medications for BD. Research Design: Participants: 30 adolescents (14-18 years old) with BD and 30 adults (19-65 years old) with BD. Measures: Blood levels of biomarkers that are associated with EMCs will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Diagnosis of BD type I, II, or NOS as determined by DSM-IV diagnostic criteria (confirmed using SCID or K-SADS)
3. Both females and males, age14 to 65 years
4. Decision by physician and patient to initiate pharmacotherapy with a traditional mood stabilizer or atypical antipsychotic
5. Able to understand and comply with requirements of the study
6. Proficient in English.

Exclusion Criteria:

1. A primary psychiatric disorder other than bipolar disorder I, II or NOS (comorbid Axis I or II disorders are permitted, as long as clinician judges that bipolar disorder is the primary condition)
2. Initiation of an antipsychotic, mood stabilizer or other medication with known endocrine-metabolic effects within 4 weeks prior to baseline visit
3. Patients who, in the investigators opinion, are unlikely to adhere to pharmacotherapy for at least 4 weeks after baseline visit
4. Significant medical condition that would contraindicate the use of mood stabilizers or atypical antipsychotics
5. Patients who are receiving pharmacological treatment for diabetes mellitus (DM), hyperlipidemia, or obesity
6. Acute or chronic medical illness (e.g. urinary tract infection, bronchitis, rheumatoid arthritis) that, as judged by the investigator, would significantly alter inflammatory, metabolic, or endocrine indices
7. Screening bloodwork that identifies any other clinically significant deviation from the reference range in clinical laboratory test results, as judged by the investigator.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Thirty adolescent participants with BD (type I, II, or not otherwise specified), and 30 adult participants with BD will be enrolled. Participants with BD will be recruited from the Youth and Adult Mood Disorder Clinics. Psychiatry Division staff will identify patients who meet the study criteria during weekly treatment team meetings. New referrals will also be screened to identify potential participants.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in metabolic syndrome components | Screening, week 4/visit 2, week 12/visit 3, week 52/final visit
  i.e. weight glucose, lipids, blood pressure, etc.

SECONDARY OUTCOMES:
Cytokines, Chemokines, Insulin, Prolactin, Thyroid Hormone | Screening, week 4/visit 2, week 12/visit 3, week 52/final visit
  * Cytokines include: pro-inflammatory markers such as c-reactive protein, interleukin-6, and tumor-necrosis factor alpha; anti-inflammatory cytokines include interleukin-4
  * Chemokines include: Leptin, Ghrelin and Adiponectin

CONTACTS AND LOCATIONS:
Overall Officials: Ayal Schaffer, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Benjamin Goldstein, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada